CLINICAL TRIAL: NCT03481530
Title: Development of Novel Predictors of Hypoglycemia for Type 2 Diabetes: Role of CGMS Usage in Predicting Risk for Hypoglycemia
Brief Title: Role of CGMS Usage in Predicting Risk for Hypoglycemia
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: MED-2017-26285
Record Dates: First submitted 2018-03-21; First posted 2018-03-29 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Type 2 Diabetes Mellitus; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Blinded: Continuing Glucose Monitoring System will be blinded
  Interventions: Device: Continuing Glucose Monitor System
- Unblinded: Continuing Glucose Monitoring System will be open. Participant can review results if they choose.
  Interventions: Device: Continuing Glucose Monitor System

INTERVENTIONS:
Device: Continuing Glucose Monitor System — glucose monitoring

SUMMARY:
This is a clinical study to examine rates hypoglycemia (self-report, EHR review, and review of values from a FDA approved continuous glucose monitoring system (CGMS)). Subjects will wear either blinded or unblinded CGMS. This is a 1:1 assignment with one group (50%) wearing 1 unblinded/1 blinded CGMS and the other group 50% wearing 2 blinded CGMS. The assignment will be computer based in a random fashion. Participants will continue with their usual diabetes management and glycemic monitoring profile as per usual. Those assigned to an unblinded CGMS can use the CGMS to manage their glucose levels at their own discretion. Individuals recruited will be those Type 2 diabetes who are deemed to be at high risk for hypoglycemia or low risk for hypoglycemia from a point score system established in an affiliated study.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes
* 18 years or older

Exclusion Criteria:

* Type 1 diabetes
* Current pregnancy or anticipation of pregnancy during study period
* At screening visit, HR> 130 or SBP>160 or DBP>100 which remains present on recheck

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with type 2 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Hypoglycemia rate | Week 16
  Overall rate

SECONDARY OUTCOMES:
Comparison hypoglycemia rate | Week 16
  Comparison between blinded and unblinded arms

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Olawsky E, Zhang Y, Eberly LE, Helgeson ES, Chow LS. A New Analysis Tool for Continuous Glucose Monitor Data. J Diabetes Sci Technol. 2022 Nov;16(6):1496-1504. doi: 10.1177/19322968211028909. Epub 2021 Jul 20. PMID 34282646